CLINICAL TRIAL: NCT02364856
Title: Assessment of Pain Through Parasympathetic Tone Analysis : Applicability in Children With Cerebral Palsy.
Brief Title: Pain Assessment in Children With Cerebral Palsy Through Parasympathetic Tone Analysis.
Status: Terminated | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Clinical Investigation Centre for Innovative Technology Network (Network); Fondation Motrice (Other)
Responsible Party: Sponsor
Other Study IDs: 2013_22; 2014-A00583-44 (Other: ID RCB number, ANSM)
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy; Pain; Children
Keywords: Autonomic Nervous System; Cerebral Palsy; Pain; Children
MeSH Terms: conditions — Cerebral Palsy; Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with cerebral palsy
  Interventions: Device: Analgesia Nociception Index

INTERVENTIONS:
Device: Analgesia Nociception Index — The Analgesia Nociception Index (ANI, MDoloris Medical Systems, Lille, France), based on Heart Rate Variability analysis, measures continuously and non-invasively the influence of Respiratory Sinus Arrhythmia on the heart rate. This 0-100 index indicates the proportion of paraS over sympathetic activity. In adults during surgery under general anesthesia, ANI decreases after painful stimulation and has been related to the balance between analgesia and nociception.
  ANI is calculated from heart rate recording.

SUMMARY:
This study evaluates Analgesia Nociception Index (Heart Rate Variability based index) and its variations after painful stimulations in children with cerebral palsy : acute procedural pain (botulinum toxin injections), and recurrent pain (physiotherapy).

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common cause of motor handicap in childhood. CP is caused by damage to the developing brain, resulting in limits in movement, posture, or communication ability. CP affects about one newborn on 450. Pain management is one of the major expectations of CP patients (La Foundation Motrice, 2009) but in this population, pain is not recognized and inadequately treated.

Autonomic nervous system (ANS) is the automatic part of our nervous system regulating vital functions like cardiac beats or respiration. It is divided in sympathetic and parasympathetic. Analysis of heart rate variability (HRV) allows isolation of variations due to parasympathetic and their study. Works from the CIC-IT 807 lead to creation of an index called ANI (Analgesia Nociception Index), which is very sensitive to pain. It is validated on adults (Jeanne, 2012). It could be helpful to assess pain in CP, particularly in patients with communication disabilities. It is important to study this new tool in CP children before developing clinical applications.

Main objective of this study is to demonstrate that ANI is relevant in CP children and that it is sensitive to pain like in adults. Population will be 40 CP children (6-18y) receiving rehabilitation therapy in specialized centres. Duration of the study is 2 years. Parent's consent should be obtained. Investigators will record heart rate of children in 3 conditions in their rehabilitation centres: usual position, acute procedural pain (botulinum toxin injections), and recurrent pain (physiotherapy). Parameters will be calculated in CIC-IT 807 lab (heart rate, ANI). Values of ANI and heart rate before and after painful stimulations will be compared. Correlation between ANI and results of usual pain assessment tools (rFLACC scale, visual analog scale) or characteristics of the population will be analyzed.

Lille University Hospital and CIC-IT 807 lab will collaborate with 2 pediatric rehabilitation centers: Centre Marc Sautelet and Zuydcoote Hospital.

Expected result is that ANI is relevant to CP children. Clinical applications are multiple: pain assessment, adaptation of medical equipment.

ELIGIBILITY:
Inclusion Criteria:

* Cerebral Palsy
* Rehabilitation care with physiotherapy and/or toxinum botulinum injections
* Absence of identified autonomic nervous system disease
* Parental and children (if applicable) consent obtained
* French National Health System cover

Exclusion Criteria:

* baseline Respiratory Frequency > 30/min
* beta-blockers or atropinic treatment
* Pacemaker, cardiac rhythm disease
* Diabetes mellitus

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Our population will be 40 CP children (6-18y) receiving rehabilitation therapy in specialized centres.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Analgesia Nociception Index ANI before and after painful stimulation | 300 seconds before and 300 seconds after painful stimulation
  ANI is calculated from heart rate recordings 300 seconds before and after painful stimulations and compared

SECONDARY OUTCOMES:
ANI at baseline | 300 seconds at rest
  ANI calculated from Heart rate recordings during 300 seconds in patient's usual position
time for recovering | 10 minutes after painful stimulation
  time for recovering baseline ANI after painful stimulation
pain score measured by Visual Analog Scale | immediately after painful stimulation
  when VAS will be applicable, children will be asked to score their pain with VAS scale; results of pain ratings with VAS will be compared to ANI results
pain score measured by rFLACC scale | immediately after painful stimulation
  rFLACC scale will be scored immediately after painful stimulation; results of pain ratings with rFLACC will be compared to ANI results
dysautonomic symptoms | inclusion
  results of ANI measures will be compared between two groups according to presence or absence of dysautonomic symptoms
Gross Motor Function Classification System | inclusion
  results of ANI measures will be compared to the severity of motor impairment through the Gross Motor Function Classification System

CONTACTS AND LOCATIONS:
Overall Officials: Justine AVEZ-COUTURIER, MD, Principal Investigator — University Hospital, Lille
Locations (3):
- France (3):
  - CHRU de Lille, Pôle Enfant, Hôpital Roger Salengro, Lille
  - Centre de Réadaptation Fonctionnelle Marc Sautelet, Villeneuve-d'Ascq
  - Hôpital maritime de Zuydcoote, Service de SSR Enfant, Zuydcoote

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeanne M, Delecroix M, De Jonckheere J, Keribedj A, Logier R, Tavernier B. Variations of the analgesia nociception index during propofol anesthesia for total knee replacement. Clin J Pain. 2014 Dec;30(12):1084-8. doi: 10.1097/AJP.0000000000000083. PMID 24525906
- [Background] Jeanne M, Clement C, De Jonckheere J, Logier R, Tavernier B. Variations of the analgesia nociception index during general anaesthesia for laparoscopic abdominal surgery. J Clin Monit Comput. 2012 Aug;26(4):289-94. doi: 10.1007/s10877-012-9354-0. Epub 2012 Mar 28. PMID 22454275
- [Background] De Jonckheere J, Rakza T, Logier R, Jeanne M, Jounwaz R, Storme L. Heart rate variability analysis for newborn infants prolonged pain assessment. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:7747-50. doi: 10.1109/IEMBS.2011.6091909. PMID 22256134
- [Background] Faye PM, De Jonckheere J, Logier R, Kuissi E, Jeanne M, Rakza T, Storme L. Newborn infant pain assessment using heart rate variability analysis. Clin J Pain. 2010 Nov-Dec;26(9):777-82. doi: 10.1097/ajp.0b013e3181ed1058. PMID 20973153